CLINICAL TRIAL: NCT04593277
Title: INSPIRE-AYA: A Multicenter Interactive Survivorship Program to Improve Healthcare Resources for Adolescent and Young Adult (AYA) Cancer Survivors
Brief Title: Interactive Survivorship Program for the Improvement of Healthcare Resources in Adolescent and Young Adult Cancer Survivors, INSPIRE-AYA Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RG1121029; NCI-2020-04792 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10470 (Other: Fred Hutch/University of Washington Cancer Consortium); U01CA246659 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage I Cutaneous Melanoma AJCC v8; Clinical Stage II Cutaneous Melanoma AJCC v8; Clinical Stage III Cutaneous Melanoma AJCC v8; Hematopoietic and Lymphoid Cell Neoplasm; Invasive Malignant Neoplasm; Leukemia; Lymphoma; Malignant Solid Neoplasm; Sarcoma; Stage I Colorectal Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Thyroid Gland Carcinoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Sarcoma; Colorectal Neoplasms; Thyroid Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (INSPIRE, telehealth care) (Experimental): Patients receive a personalized SCP and use the INSPIRE mobile application. Patients may receive telehealth stepped care after 1 month.
  Interventions: Other: Internet Mobile Technology; Other: Questionnaire Administration; Procedure: Supportive Care; Other: Informational Intervention
- Arm II (control website) (Active Comparator): Patients receive access to a study-specific control website that has annotated links to existing resources for AYA survivors. After 12 months, patients receive a personalized SCP and have access to the digital INSPIRE intervention program without telehealth calls.
  Interventions: Other: Internet-Based Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet Mobile Technology — Use INSPIRE mobile application
  Other Names: www-mobile
  Arms: Arm I (INSPIRE, telehealth care)
Other: Internet-Based Intervention — Access to a study-specific control website
  Arms: Arm II (control website)
Other: Questionnaire Administration — Ancillary studies
Procedure: Supportive Care — Receive telehealth stepped care
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Arm I (INSPIRE, telehealth care)
Other: Informational Intervention — Receive printed SCP materials
  Arms: Arm I (INSPIRE, telehealth care)

SUMMARY:
This trial studies how well an interactive survivorship program works in improving healthcare resources in adolescent and young adult cancer survivors. By improving access to survivorship resources, health literacy, self-management skills, and support, an interactive survivorship program may help to improve adherence to adolescent and young adult healthcare guidelines and reduce cancer-related distress.

DETAILED DESCRIPTION:
OUTLINE: Patients who have one or more elevated distress or low cardiometabolic or cancer health care adherence are randomized to Arm I or II.

ARM I (INTERVENTION): Patients receive a personalized Survivorship Care Plan (SCP) and use the Interactive Survivorship Program to Improve Healthcare Resources (INSPIRE) mobile application. Patients may receive telehealth stepped care after 1 month.

ARM II (CONTROL): Patients receive access to a study-specific control website that has annotated links to existing resources for adolescent and young adult (AYA) survivors. After 12 months, patients receive a personalized SCP and have access to the digital INSPIRE intervention program without telehealth calls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a first invasive malignancy of leukemia, lymphoma, melanoma, sarcoma, breast, thyroid, or colorectal cancer (stage 1-3 for solid tumors) between the ages of 15-39 years
* Current age >= 18 when approached
* Currently within 1 to 5 years from the time of diagnosis
* Completed active treatment for disease >= 6 months previously
* Received a therapeutic intervention (with curative intent if advanced stage disease) that included any of the following modalities: surgery, cytotoxic chemotherapy, biological or targeted agents, radiation therapy
* English proficiency adequate to complete assessments
* Access to email and smartphone mobile app and or internet

Exclusion Criteria:

* Diagnosed with a subsequent invasive malignancy other than non-melanoma skin cancer
* Received hematopoietic stem cell transplant
* Health issues prohibiting computer use or ability to comply with study procedures
* Residing in an institution or other living situation where health care decisions are not made by the participant (e.g., hospitalized, prisoners, living in a rehabilitation facility)
* Does not complete baseline patient reported outcome (PRO) assessment items required to determine stratification or whether the survivor meets inclusion and exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2022-10-23 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change in distress score from baseline to 3 months | From baseline to 3 months
  Will be assessed by Cancer and Treatment Distress (CTXD). The CTXD is a 22 item Likert type scale that contains 6 subscales: uncertainty, health burden, identity, medical demands, finances, and family strain. Scores on individual items range from 0 (none) to 3 (severe) distress related to an aspect of the cancer experience. Patients will meet the primary endpoint for lack of distress if they score < 0.9 on the CTXD.
Change in distress score from baseline to 12 months | From baseline to 12 months
  Will be assessed by Cancer and Treatment Distress (CTXD). The CTXD is a 22 item Likert type scale that contains 6 subscales: uncertainty, health burden, identity, medical demands, finances, and family strain. Scores on individual items range from 0 (none) to 3 (severe) distress related to an aspect of the cancer experience. Patients will meet the primary endpoint for lack of distress if they score < 0.9 on the CTXD.

SECONDARY OUTCOMES:
Proportion of healthcare adherence (HCA)-all | At 12 months
  Patients will meet HCA endpoint if their percent of recommended screenings obtained within the past 12 months is >= 80% for HCA-all.
Proportion of HCA-cardiometabolic surveillance (CM) | At 12 months
  Patients will meet each HCA endpoint if their percent of recommended screenings obtained within the past 12 months is >= 80% for HCA-CM.
Proportion of HCA-cancer surveillance (SM) | At 12 months
  Patients will meet each HCA endpoint if their percent of recommended screenings obtained within the past 12 months is >= 80% for HCA-SM.

CONTACTS AND LOCATIONS:
Overall Officials: K. Scott Baker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (5):
- United States (5):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT04593277/ICF_000.pdf